CLINICAL TRIAL: NCT00760214
Title: A Double-Blind, Randomized, Parallel-Group Study to Compare the Efficacy and Safety of TAK-491 With Ramipril in Subjects With Essential Hypertension
Brief Title: Efficacy and Safety Study of Azilsartan Medoxomil Compared to Ramipril for Treating Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-491-020; 2007-002583-10 (EudraCT Number); U1111-1113-8982 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-24; First posted 2008-09-26 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Hypertension; Drug Therapy; Blood Pressure, High; Vascular Disease; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Essential Hypertension; Vascular Diseases; Cardiovascular Diseases | interventions — azilsartan medoxomil; azilsartan; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Ramipril 10 mg QD (Active Comparator)
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Azilsartan medoxomil — Azilsartan medoxomil 20 mg, tablets, orally, once daily for two weeks; then increased to 40 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 20 mg, tablets, orally, once daily for two weeks; then increased to 80 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Ramipril — Ramipril 2.5 mg, tablets, orally, once daily for two weeks; then increased to 10 mg, tablets, orally, once daily for up to 22 weeks.
  Other Names: Tritace; Ramace; Altace
  Arms: Ramipril 10 mg QD

SUMMARY:
The purpose of this study is to determine the efficacy and safety of azilsartan medoxomil, once daily (QD), compared to ramipril for treating Essential Hypertension.

DETAILED DESCRIPTION:
A major component of blood pressure regulation is the renin-angiotensin-aldosterone system, a system of hormone-mediated feedback interactions that results in the relaxation or constriction of blood vessels in response to various stimuli. Angiotensin II, a polypeptide hormone, is formed from angiotensin I in a reaction catalyzed by angiotensin-converting enzyme as part of the renin-angiotensin-aldosterone system. Angiotensin II is the principal pressor agent of the renin-angiotensin-aldosterone system with a myriad of effects on the cardiovascular system and on electrolyte homeostasis. Two receptors for angiotensin II have been identified. Angiotensin II type 1 receptors are located predominantly in vascular smooth muscle, where activation by angiotensin II results in vasoconstriction, hypertrophic proliferation, and inflammation. In contrast, stimulation of angiotensin II type 2 receptors by angiotensin II results in vasodilatation, antiproliferative effects that are opposite from those of angiotensin II type 1 receptor stimulation.

Drugs that modulate the renin-angiotensin-aldosterone system are used commonly worldwide for the treatment of hypertension. Of these, some block the synthesis of angiotensin II by inhibiting angiotensin-converting enzymes, while others inhibit the action of angiotensin II by binding directly to the angiotensin II type 1 receptor (called angiotensin II receptor blockers), thereby causing vasodilatation of blood vessels, resulting in a reduction in blood pressure. The effects of angiotensin II receptor blockers on other conditions in which the renin-angiotensin-aldosterone system plays a significant role, such as congestive heart failure, postmyocardial infarction management and diabetic nephropathy have also been investigated.

Although antihypertensive agents are effective at the appropriate dose, the majority have side effects that limit their use. Angiotensin-converting enzyme inhibitors are commonly associated with cough and more rarely with angioedema. Beta-blockers are associated with fatigue and erectile dysfunction, calcium antagonists with peripheral edema and diuretics with metabolic complications. As a class, angiotensin II receptor blockers generally are considered more tolerable than other classes of hypertensive agents, although there is still a need for compounds with improved tolerability and efficacy for the treatment of hypertension.

TAK-491 (azilsartan medoxomil) is an angiotensin II receptor blocker with high affinity for, and selective antagonistic activity at, the angiotensin II type 1 receptor, and is being developed for clinical use as an antihypertensive agent.

Ramipril is an angiotensin-converting enzyme inhibitor widely prescribed in Europe and Asia for the treatment of mild to moderate essential hypertension.

This study is designed to compare the efficacy and safety/tolerability of azilsartan medoxomil and ramipril for the treatment of hypertension.

Participants in this study will be seen twice during the first month, then once a month for five months. Participants will also be required to fast for 8 hours prior to each visit to the study center. Total duration of study participation is 24-weeks, plus a safety follow up phone call after the study has ended.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertension (sitting systolic blood pressure between 150 and 180 mm Hg, inclusive).
2. A female participant of childbearing potential who is sexually active agrees to use adequate contraception from screening throughout the duration of the study, and cannot be pregnant.
3. Has clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) within the reference range for the testing laboratory at Screening or the results are deemed not clinically significant for inclusion into this study by the investigator.
4. Is willing to discontinue current antihypertensive medications at Screening Day -21. If the participant is on amlodipine prior to screening, the participant is willing to discontinue this medication at Screening Day -28.

Exclusion Criteria:

1. Has an systolic blood pressure greater than 180 mmHg or diastolic blood pressure greater than 114 mmHg at Randomization.
2. Is taking or expected to take an excluded medication including antihypertensive agents, insulin or other agents that alter blood pressure.
3. Is hypersensitive to angiotensin II receptor blockers and/or angiotensin-converting enzyme inhibitors.
4. Has a recent history within the last 6 months of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Has clinically significant cardiac conduction defects (eg, third-degree atrioventricular block, left bundle branch block, sick sinus syndrome, atrial fibrillation or flutter).
6. Has hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
7. Has secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
8. Is noncompliant (less than 70% or greater than 130%) with study medication during placebo run-in period.
9. Has severe renal dysfunction or disease (based on calculated creatinine clearance less than 30 mL/min/1.73 m² at Screening).
10. Has known or suspected unilateral or bilateral renal artery stenosis.
11. Has a history of drug or alcohol abuse within the past 2 years.
12. Has a previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug. (This criterion does not apply to those participants with basal cell or stage I squamous cell carcinoma of the skin).
13. Has type 1 or poorly controlled type 2 diabetes mellitus (hemoglobin A1c greater than 8.0%) or is taking insulin.
14. Has hyperkalemia as defined by the central laboratory normal reference range at Screening.
15. Has an upper arm circumference less than 24 cm or greater than 42 cm.
16. Works night (third) shift (defined as 11 PM to 7 AM).
17. Has an alanine aminotransferase level at Screening of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
18. Is currently participating in another investigational study or has participated in an investigational study within 30 days prior to Screening.
19. Has any other serious disease or condition at Screening or Randomization that would compromise participant's safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
20. Has been randomized in a previous azilsartan medoxomil study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda Global Research & Development Center (Europe), Ltd.
Locations (72):
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Estonia (4):
  - Paide
  - Tallinn
  - Tartu
  - Viljandi
- Finland (4):
  - Joensuu
  - Mikkeli
  - Tampere
  - Turku
- Germany (20):
  - Augsburg
  - Bad Krozingen
  - Bad Segeberg
  - Berlin
  - Cologne
  - Dortmund
  - Dresden
  - Essen
  - Frankfurt
  - Goch
  - Großheirath
  - Hamburg
  - Karlsruhe
  - Künzing
  - Leipzig
  - Lübeck
  - Mannheim
  - München
  - Nuremberg
  - Siegen
- Netherlands (9):
  - Deurne
  - Ewijk
  - Geleen
  - Lichtenvoorde
  - Oude Pekela
  - Rijswijk
  - Roelofarendsveen
  - Rotterdam
  - Wildervank
- Poland (11):
  - Gdansk
  - Gniewkowo
  - Kamieniec Ząbkowicki
  - Katowice
  - Libiąż
  - Lodz
  - Oława
  - Poznan
  - Płock
  - Skierniewice
  - Tarnów
- Russia (3):
  - Moscow
  - Perm
  - Saint Petersburg
- Serbia (4):
  - Belgrade
  - Niš
  - Niška Banja
  - Zemun
- Slovakia (5):
  - Bratislava
  - Galanta
  - Levice
  - Lučenec
  - Rimavská Sobota
- Sweden (7):
  - Boden
  - Gothenburg
  - Luleå
  - Lund
  - Malmo
  - Örebro
  - Skene

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 122 investigative sites in Bulgaria, Estonia, Finland, Germany, the Netherlands, Poland, Russia, Serbia and Montenegro, Slovakia and Sweden from 24 January 2008 to 21 April 2009.
Pre-assignment Details: Participants with essential hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for two weeks; then increased to 40 mg, tablets, orally, once daily for up to 22 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 20 mg, tablets, orally, once daily for two weeks; then increased to 80 mg, tablets, orally, once daily for up to 22 weeks.
- Ramipril 10 mg QD: Ramipril 2.5 mg, tablets, orally, once daily for two weeks; then increased to 10 mg, tablets, orally, once daily for up to 22 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Started | 295 | 294 | 296
Completed | 265 | 264 | 255
Not Completed | 30 | 30 | 41
Not completed — Adverse Event | 8 | 9 | 12
Not completed — Protocol Violation | 3 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 12 | 14 | 13
Not completed — Lack of Efficacy | 3 | 2 | 4
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Other | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD | Total
Number analyzed (Participants) | 295 | 294 | 295 | 884
Age, Customized [Number; unit: Participants]
  <45 years | 40 | 45 | 30 | 115
  Between 45 and 64 years | 166 | 168 | 195 | 529
  ≥65 years | 89 | 81 | 70 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 136 | 149 | 421
  Male | 159 | 158 | 146 | 463

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure.
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 24 relative to baseline. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 291 | 289 | 290
mmHg | -20.63 (0.946) | -21.24 (0.949) | -12.22 (0.948)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value presented. Overall 0.05 level of significance for multiple comparisons controlled using stepwise testing procedure; Mean Difference (Final Values) = -8.41, 95% CI 2-sided [-11.04 to -5.78]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.03, 95% CI 2-sided [-11.66 to -6.39]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 24 relative to baseline. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 24.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 291 | 289 | 290
mmHg | -10.18 (0.553) | -10.54 (0.556) | -4.87 (0.555)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value presented; Mean Difference (Final Values) = -5.31, 95% CI 2-sided [-6.85 to -3.78]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.66, 95% CI 2-sided [-7.21 to -4.12]

3. Secondary Outcome: Change From Baseline in 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -12.65 (1.006) | -12.29 (0.992) | -7.83 (1.022)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.82, 95% CI 2-sided [-7.64 to -2.01]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.47, 95% CI 2-sided [-7.27 to -1.66]

4. Secondary Outcome: Change From Baseline in 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -8.03 (0.655) | -8.32 (0.646) | -5.26 (0.666)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-4.61 to -0.94]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.06, 95% CI 2-sided [-4.89 to -1.24]

5. Secondary Outcome: Change From Baseline in the 12-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -12.06 (1.103) | -11.71 (1.087) | -8.28 (1.121)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.77, 95% CI 2-sided [-6.87 to -0.68]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.029, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.43, 95% CI 2-sided [-6.50 to -0.36]

6. Secondary Outcome: Change From Baseline in the 12-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring
Description: The change in the 12-hour mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -7.71 (0.743) | -8.07 (0.732) | -5.65 (0.755)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.052, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.06, 95% CI 2-sided [-4.15 to 0.02]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.022, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.42, 95% CI 2-sided [-4.49 to -0.35]

7. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -12.61 (1.047) | -12.35 (1.032) | -8.08 (1.064)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.53, 95% CI 2-sided [-7.46 to -1.59]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -4.26, 95% CI 2-sided [-7.18 to -1.35]

8. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 8 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 131 | 135 | 127
mmHg | -8.19 (0.700) | -8.53 (0.689) | -5.55 (0.711)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.64, 95% CI 2-sided [-4.60 to -0.68]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -2.98, 95% CI 2-sided [-4.93 to -1.04]

9. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 130 | 135 | 127
mmHg | -12.82 (1.135) | -12.69 (1.115) | -6.87 (1.147)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.95, 95% CI 2-sided [-9.12 to -2.77]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.82, 95% CI 2-sided [-8.96 to -2.67]

10. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 130 | 135 | 127
mmHg | -7.44 (0.764) | -8.20 (0.750) | -4.43 (0.773)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-5.15 to -0.88]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -3.77, 95% CI 2-sided [-5.89 to -1.65]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 130 | 135 | 127
mmHg | -15.60 (1.172) | -14.93 (1.151) | -6.73 (1.186)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -8.87, 95% CI 2-sided [-12.15 to -5.60]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -8.20, 95% CI 2-sided [-11.46 to -4.95]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 24 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 24.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Number analyzed (Participants) | 130 | 135 | 127
mmHg | -10.21 (0.898) | -9.85 (0.883) | -4.53 (0.909)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.68, 95% CI 2-sided [-8.19 to -3.17]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Ramipril 10 mg QD; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = -5.32, 95% CI 2-sided [-7.81 to -2.82]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Ramipril 10 mg QD
Serious Adverse Events (participants affected / at risk) | 8/294 | 12/293 | 6/293
Other Adverse Events (participants affected / at risk) | 22/294 | 16/293 | 36/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=294) | Azilsartan Medoxomil 80 mg QD (N=293) | Ramipril 10 mg QD (N=293)
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=294) | Azilsartan Medoxomil 80 mg QD (N=293) | Ramipril 10 mg QD (N=293)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 24
Nasopharyngitis (Infections and infestations) | 19 | 13 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.